CLINICAL TRIAL: NCT06705699
Title: Urethral Mobilisation Versus Mathieu Technique for Repair of Distal Hypospadias
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Elnoby Mohamed Abdelhameed, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Treatment of Hypospadias
Record Dates: First submitted 2024-11-20; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Hypospadias Repair Surgery
Keywords: mathieu; urethral; mobilisation; hypospadias
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Who Masked: Participant
Masking Description: data analyst
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urethral Mobilization Technique (Experimental): • Description: Involves mobilizing the urethral tube proximally and advancing it distally to the glans. The urethra is repositioned and sutured at the neomeatal position.
  Interventions: Procedure: Urethral mobilisation
- Mathieu Technique (Experimental): • Description: Utilizes a perimeatal-based flap, which is flipped up to create the neourethra.
  Interventions: Procedure: Mathieu

INTERVENTIONS:
Procedure: Urethral mobilisation — Involves mobilizing the urethral tube proximally and advancing it distally to the glans. The urethra is repositioned and sutured at the neomeatal position.
  Arms: Urethral Mobilization Technique
Procedure: Mathieu — Utilizes a perimeatal-based flap, which is flipped up to create the neourethra.
  Arms: Mathieu Technique

SUMMARY:
The aim of this research is to compare the surgical outcomes of urethral mobilization and the Mathieu technique in treating distal penile hypospadias. The study will evaluate complication rates such as fistula formation and meatal stenosis, assess functional outcomes related to urinary stream quality, and analyze cosmetic results including the appearance of the neomeatus. Ultimately, the goal is to provide evidence-based guidance for choosing the most appropriate technique to optimize surgical outcomes and patient satisfaction.

DETAILED DESCRIPTION:
Hypospadias is a common congenital malformation of the male genitalia, characterized by the abnormal positioning of the urethral meatus along the ventral surface of the penis . It affects approximately 1 in every 200 male births and is most frequently observed in its distal form, where the urethral opening is located near the glans . Surgical correction of hypospadias is necessary to ensure proper urinary function, achieve a cosmetically acceptable appearance, and prevent future complications such as chordee or abnormal curvature of the penis . There are several surgical techniques available for repairing distal penile hypospadias, each with its own advantages and drawbacks. Among these, the Mathieu technique and the urethral mobilization technique are two commonly employed approaches.

The Mathieu technique, first introduced in 1932, uses a perimeatal-based flap to reconstruct the urethra. It is a reliable and well-established method that is associated with a relatively low rate of complications, such as urethrocutaneous fistula and meatal stenosis. However, one of the main limitations of the Mathieu technique is the creation of a rounded or horizontal meatus, which is often considered less cosmetically pleasing compared to the more natural slit-like meatus formed by other techniques. Despite this drawback, the Mathieu technique remains a popular choice for surgeons, particularly in cases where the urethral plate is well-developed and no additional ventral curvature correction is required.

The urethral mobilization technique, on the other hand, involves the proximal mobilization and distal advancement of the native urethra to the tip of the glans without using a preputial flap. This approach can be especially beneficial for boys who have already undergone circumcision, as it does not rely on the availability of a preputial skin flap. Studies suggest that urethral mobilization results in satisfactory functional outcomes and a lower incidence of certain complications, such as meatal stenosis and postoperative fistula formation. Furthermore, it is considered a straightforward procedure that avoids extensive tissue dissection, making it an appealing option for selected cases of distal hypospadias.

While both techniques have demonstrated satisfactory outcomes, there is a need for a comprehensive comparison to evaluate their effectiveness and safety profiles. Existing literature suggests that urethral mobilization results in lower complication rates compared to the Mathieu technique in specific clinical settings. Additionally, a study by reported that the Mathieu technique with an incision of the urethral plate showed significantly fewer complications, including meatal stenosis and fistula formation, compared to the tubularized incised-plate (TIP) technique, further demonstrating the variability in outcomes based on surgical approach.

ELIGIBILITY:
Inclusion Criteria:• Male patients aged 6 months to 7 years.

* Diagnosed with distal penile hypospadias (coronal, or subcoronal types).
* Mild to no chordee present (curvature <30°).
* No associated with severe genital anomalies.

Exclusion Criteria:

* Patients with proximal hypospadias (midshaft, penoscrotal, or perineal).

  * Presence of significant chordee requiring separate corrective procedures.
  * Hypoplastic or poorly developed urethral plate that is unsuitable for surgical repair.
  * Previous hypospadias repair surgery.
  * Patients with severe comorbidities or conditions that could increase the risk of surgery (e.g., severe cardiac anomalies).

Ages: 6 Months to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — male children with hypospadias
Enrollment: 60 (Estimated)
Dates: Start 2024-11-25 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
urethrocutaneous fistula | 1 month
  Absence of urethrocutaneous fistula formation
  • Postoperative complication rates, including urethrocutaneous fistula formation, meatal stenosis, wound infection, hematoma, and retraction of the neomeatus.
meatal stenosis | 2 months
  absence of meatal stenosis
wound infection | 1 week
  absence of wound infection
hematoma | 3 days
  absence of hematoma
neomeatus retraction | 3 months
  absence of retraction of the neomeatus.

SECONDARY OUTCOMES:
quality of the urinary stream | 2 months
  Functional outcomes assessed by the quality of the urinary stream (single stream, narrow stream, sprayed stream).
cosmetic | 3 months
  Cosmetic outcomes evaluated using the HOSE scoring system to assess the appearance.
shape | 3 months
  Cosmetic outcomes evaluated using the HOSE scoring system to assess the shape.
position of the neomeatus | 3 months
  Cosmetic outcomes evaluated using the HOSE scoring system to assess the position of the neomeatus.

CONTACTS AND LOCATIONS:
Overall Officials: ibrahim farag, prof, Study Director — Assiut University; tarek hassan, prof, Study Director — assuit

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Martínez ADCR, Barrientos-Villegas S, Mondragón CFM, Hernández EF, Martínez-Sosa IP, Mera BB, et al. Hypospadias: a review. International Surgery Journal. 2024;11(8):1439.